CLINICAL TRIAL: NCT00590889
Title: Artificial Valve Endocarditis Reduction Trial
Acronym: AVERT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: A post-PMA begun in 1998; enrollment halted in 2000 due to an anomaly in one study arm. The protocol required annual study visits after 2000.
Sponsor: Abbott Medical Devices (Industry)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 979
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Results first posted 2015-12-22 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Aortic Valve Disease; Mitral Valve Disease; Endocarditis
Keywords: artificial heart valve; mitral heart valve; aortic heart valve; endocarditis; Aortic valve disease requiring replacement; Mitral valve disease requiring replacement
MeSH Terms: conditions — Aortic Valve Disease; Endocarditis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- St. Jude Medical (SJM) Conventional (Other): St. Jude Medical (SJM) Standard Masters Series Mechanical Heart Valve with Conventional Cuff
  Interventions: Device: Artificial Mechanical Heart Valve
- St. Jude Medical (SJM) Silzone (Other): St. Jude Medical (SJM) Masters Series Mechanical Heart Valve with Silzone Coating
  Interventions: Device: Artificial Mechanical Heart Valve

INTERVENTIONS:
Device: Artificial Mechanical Heart Valve — Both arms used market released mechanical heart valves in accordance with approved labeling

SUMMARY:
The purpose of this study is to investigate whether the Silzone coated sewing cuff reduces the incidence of prosthetic valve endocarditis (PVE).

DETAILED DESCRIPTION:
The purpose of this study is to investigate whether the Silzone coated sewing cuff reduces the incidence of prosthetic valve endocarditis. The null and alternative hypotheses of this study are:

* Ho: Patients receiving SJM Masters Series valves with Silzone coating will have an equal incidence of PVE when compared to those receiving the conventional cuff.
* Ha: Patients receiving SJM Masters Series valves with Silzone coating will have a reduced incidence of PVE when compared to those receiving the conventional cuff.

ELIGIBILITY:
Inclusion Criteria:

* The patient requires an isolated mitral, isolated aortic, or double (aortic and mitral) valve replacement
* The patient is a candidate to receive an SJM (St. Jude Medical) Masters Series valve(s) with either the conventional cuff or the cuff with Silzone coating
* The patient (or legal guardian) has signed a study-specific consent form agreeing to the randomization, data collection, and follow-up requirements

Exclusion Criteria:

* The patient has a medical condition which contraindicates implantation of the SJM Masters Series with Silzone coating
* The patient already has a prosthetic valve other than the valve being replaced at this time
* The patient requires a tricuspid valve replacement

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 807 (Actual)
Dates: Start 1998-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (7):
  - Florida Heart Group, Orlando, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Womens Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Sisters of Providence Health System, Portland, Oregon
  - Texas Heart Institute, Houston, Texas
  - LDS Hospital, Salt Lake City, Utah
- Canada (2):
  - University of Alberta Hospital, Edmonton, Alberta
  - University of British Columbia, Vancouver, British Columbia
- Hôpital G. Et R. Laënnec, Nantes, France
- Deutches Herzzentrum Berlin, Berlin, Germany
- Fond Ne Centro S. Raffaele, Milan, Italy
- St. Antonius Ziekenhuis, Nieuwegein, Netherlands
- Hospital 12 de Octubre, Madrid, Spain
- Switzerland (2):
  - Inselspital, Bern
  - Hopital Regional-Service de Cardiologie, Sion

REFERENCES:
- [Background] Schaff H, Carrel T, Steckelberg JM, Grunkemeier GL, Holubkov R. Artificial Valve Endocarditis Reduction Trial (AVERT): protocol of a multicenter randomized trial. J Heart Valve Dis. 1999 Mar;8(2):131-9. PMID 10224570
- [Result] Davila-Roman VG, Waggoner AD, Kennard ED, Holubkov R, Jamieson WR, Englberger L, Carrel TP, Schaff HV; Artificial Valve Endocarditis Reduction Trial echocardiography study. Prevalence and severity of paravalvular regurgitation in the Artificial Valve Endocarditis Reduction Trial (AVERT) echocardiography study. J Am Coll Cardiol. 2004 Oct 6;44(7):1467-72. doi: 10.1016/j.jacc.2003.12.060. PMID 15464329
- [Result] Schaff HV, Carrel TP, Jamieson WR, Jones KW, Rufilanchas JJ, Cooley DA, Hetzer R, Stumpe F, Duveau D, Moseley P, van Boven WJ, Grunkemeier GL, Kennard ED, Holubkov R; Artificial Valve Endocarditis Reduction Trial. Paravalvular leak and other events in silzone-coated mechanical heart valves: a report from AVERT. Ann Thorac Surg. 2002 Mar;73(3):785-92. doi: 10.1016/s0003-4975(01)03442-7. PMID 11899956
- [Result] Englberger L, Carrel T, Schaff HV, Kennard ED, Holubkov R; AVERT Investigators. Differences in heart valve procedures between North American and European centers: a report from the Artificial Valve Endocarditis Reduction Trial (AVERT). J Heart Valve Dis. 2001 Sep;10(5):562-71. PMID 11603594
- [Result] Englberger L, Schaff HV, Jamieson WR, Kennard ED, Im KA, Holubkov R, Carrel TP; AVERT Investigators. Importance of implant technique on risk of major paravalvular leak (PVL) after St. Jude mechanical heart valve replacement: a report from the Artificial Valve Endocarditis Reduction Trial (AVERT). Eur J Cardiothorac Surg. 2005 Dec;28(6):838-43. doi: 10.1016/j.ejcts.2005.09.014. Epub 2005 Nov 7. PMID 16275007

RESULTS

PARTICIPANT FLOW:
Groups:
- SJM Conventional: SJM Standard Masters Series Mechanical Heart Valve with Conventional Cuff
  Artificial Mechanical Heart Valve: Both arms used market released mechanical heart valves in accordance with approved labeling
- SJM Silzone: SJM Masters Series Mechanical Heart Valve with Silzone Coating
  Artificial Mechanical Heart Valve: Both arms used market released mechanical heart valves in accordance with approved labeling
Period: Overall Study
Arm/Group | SJM Conventional | SJM Silzone
Started | 404 | 403
Completed | 118 | 104
Not Completed | 286 | 299

BASELINE CHARACTERISTICS:
Population: 1 subject age is missing
Groups:
- Total: Total of all reporting groups
Arm/Group | SJM Conventional | SJM Silzone | Total
Number analyzed (Participants) | 404 | 403 | 807
Age, Customized [Number; unit: participants] — We are missing 1 person's age in the Conventional group which would make the total 404
  participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 244 | 218 | 462
    >=65 years | 159 | 185 | 344
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 168 | 165 | 333
  Male | 236 | 238 | 474

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Prosthetic Valve Endocarditis Comparing Conventional Valves to Silzone™ Coated Valves.
Description: Patient response to treatment with the Silzone™ treated valve will be evaluated based upon the incidence of early and late PVE (prosthetic valve endocarditis) in the treatment group vs. the control group.
Time Frame: 1 year
Population: subjects randomized into the study
Measure: Number; unit: participants
Arm/Group | SJM Conventional | SJM Silzone
Number analyzed (Participants) | 404 | 403
participants | 10 | 9

ADVERSE EVENTS:
Time Frame: 12 years
Groups:
- Adverse Events for the Conventional Group: These patients received a conventional heart valve.
- Adverse Events for the Silzone™ Group: These patients received the Silzone™ treated heart valve.
Arm/Group | Adverse Events for the Conventional Group | Adverse Events for the Silzone™ Group
Serious Adverse Events (participants affected / at risk) | 194/404 | 261/403
Other Adverse Events (participants affected / at risk) | 124/404 | 118/403
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adverse Events for the Conventional Group (N=404) | Adverse Events for the Silzone™ Group (N=403)
Explant due to PV (para-valvular) leak (Cardiac disorders) | 3 (3) | 16 (16)
All reported explants (Cardiac disorders) | 11 (11) | 27 (27)
All reported explants/repairs (Cardiac disorders) | 16 (16) | 33 (33)
Major PV (Para-Valvular) leak (Cardiac disorders) | 7 (7) | 19 (19)
Stroke/RIND (Cardiac disorders) | 27 (27) | 26 (26)
All Cause Mortality (Cardiac disorders) | 130 (130) | 140 (140)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adverse Events for the Conventional Group (N=404) | Adverse Events for the Silzone™ Group (N=403)
Confirmed TE (Cardiac disorders) | 61 (61) | 59 (59)
Confirmed TE without TIA (Cardiac disorders) | 35 (35) | 32 (32)
Confimred TE Stroke (Cardiac disorders) | 18 (18) | 18 (18)
Endocarditis (Cardiac disorders) | 10 (10) | 9 (9)

LIMITATIONS AND CAVEATS:
This study was terminated early. No final report was created.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No